Conservative Management Equally Effective to New Suture Anchor Technique for Acute Mallet Finger Deformity: A Prospective Randomized Clinical Trial

Date: May 23th, 2013

## **Statistical Analysis**

Quantitative variables are described as means and standard deviations or medians and interquartile range. Fisher's exact or the Mann-Whitney U test (asymmetric distribution) was applied to compare the two groups in relation to the quantitative outcomes. RO M value was analyzed using OpenEpi, a Windows-based software program. The level of significance was set at 5%, where P < 0.05 was considered statistically significant.